CLINICAL TRIAL: NCT04049175
Title: A 52 Week, Randomised, Double Blind, Multinational, Multicentre, 4-arm Parallel Group Trial to Assess the Efficacy and Safety of 3 Doses of CHF 6532 Compared to Placebo on Top of Standard of Care in Patients With Uncontrolled Severe Eosinophilic Asthma
Brief Title: Efficacy and Safety of CHF 6532 in Patients With Uncontrolled Severe Eosinophilic Asthma
Acronym: PERSEA
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: An interim analysis run by an independent data monitoring committee (DMC) to assess futility met the protocol-defined futility rules. The DMC recommended to stop the study for futility. The Sponsor issued a notification of early study termination.
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLI-06532AA1-01; 2018-003548-22 (EudraCT Number)
Record Dates: First submitted 2019-08-05; First posted 2019-08-08 (Actual); Last update posted 2022-04-08 (Actual); Status verified 2022-03

CONDITIONS: Asthma; Eosinophilic
MeSH Terms: conditions — Pulmonary Eosinophilia

STUDY DESIGN:
Intervention Model Description: Placebo controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Treatment A (Experimental): Administration of CHF 6532 Dose #1
  Interventions: Drug: Treatment A
- Treatment B (Experimental): Administration of CHF 6532 Dose #2
  Interventions: Drug: Treatment B
- Treatment C (Experimental): Administration of CHF 6532 Dose #3
  Interventions: Drug: Treatment C
- Treatment D (Placebo Comparator): Administration of CHF 6532 Placebo
  Interventions: Drug: Treatment D

INTERVENTIONS:
Drug: Treatment A — Tablet of CHF 6532
  Other Names: CHF 6532
  Arms: Treatment A
Drug: Treatment B — Tablet of CHF 6532
  Other Names: CHF 6532
  Arms: Treatment B
Drug: Treatment C — Tablet of CHF 6532
  Other Names: CHF 6532
  Arms: Treatment C
Drug: Treatment D — Tablet of CHF 6532 placebo
  Other Names: CHF 6532
  Arms: Treatment D

SUMMARY:
The purpose of this phase III Study is to demonstrate the efficacy of at least one dose of CHF 6532 on moderate and severe asthma exacerbations rate compared to placebo.

DETAILED DESCRIPTION:
This is a phase III, randomised, double-blind, placebo controlled multinational, multicentre, 4-arm parallel-group, study evaluating 3 doses of CHF 6532.

The effect of CHF 6532 compared to Placebo on severe asthma exacerbations over 52 weeks of treatment will be assessed.

The effect of CHF 6532 compared to Placebo in terms of change from baseline in pre-dose morning Forced Expiratory Volume in the first second (FEV1) as well as on St. George's Respiratory Questionnaire (SGRQ), Asthma Control Questionnaire (ACQ-5) and Asthma Quality of Life Questionnaire (AQLQ+12), at Week 52 will be assessed .

The inter-subject variability in the drug exposure and the effect of selected covariates on Pharmacokinetics (PK) will be investigated.

The impact of study treatments on health economics outcomes will be also investigated.

Standard safety assessments will be conducted during the Study, including electrocardiograms (ECGs), vital signs and laboratory tests.

Approximately 1392 severe eosinophilic asthmatic adult subjects and additional 248 severe eosinophilic asthmatic adolescent subjects will be randomised in about 150 investigational sites.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged ≥12 years and ≤75 years with a diagnosis of asthma [according to Global Initiative for Asthma (GINA)] for a period of at least 24 months prior to screening.
* Subjects treated according to GINA step 4/5 with stable high-dose inhaled corticosteroids (ICS) plus a long-acting β2 agonist (LABA)
* 2 Asthma exacerbations history.
* A positive response to a reversibility test at screening.
* Subjects with evidenced eosinophilic airway inflammation at screening visit.
* Subjects with uncontrolled asthma as evidenced by ACQ-5 score ≥1.5 at screening and randomisation visits.
* Subjects with co-operative attitude and ability to perform all trial related procedures.
* Ability of patient to swallow tablets.

Exclusion Criteria:

* Pregnant or lactating women and all women of childbearing potential unless are using a highly effective birth control method.
* Run-in compliance < 50% at randomisation
* Hospitalisation, emergency room admission or use of systemic corticosteroids for an asthma exacerbation or respiratory tract infection in the 4 weeks prior to screening visit or during the run-in period.
* Subjects with a history of near fatal asthma or of a past hospitalisation for asthma in intensive care unit which, in the judgement of the investigator, may place the subjects at undue risk.
* Subjects with a history of more than 2 episodes of confirmed bacterial lower respiratory tract infection within the year prior to screening or with a bacterial lower respiratory tract infection during the run-in.
* History of diagnosis of Chronic Obstructive Pulmonary Disease (COPD), cystic fibrosis, bronchiectasis or alpha-1 antitrypsin deficiency, or any other significant lung disease which may interfere with study evaluations.
* Subjects with a marked resting baseline prolongation of mean QTc interval.
* Subjects with a family history of long QT Syndrome.
* Subjects with hypokalemia at screening.
* Subjects who have known clinically significant cardiovascular conditions.
* Subjects with a history of symptoms or significant neurological disease.
* Subjects with clinically significant abnormal serum biochemistry, haematology (not associated with the study indication) at screening according to the investigators judgement.
* Current smokers or ex-smokers with total cumulative exposure ≥10 pack-years or having stopped smoking less than one year prior to screening visit.
* Subjects with historical or current evidence of uncontrolled concurrent disease.
* Subjects with a history of hypersensitivity and/or idiosyncrasy to any of the test compounds or excipients employed in this study.
* Subjects receiving treatment with any drug known to have a well-defined potential for hepatotoxicity within the previous 3 months before the screening visit.
* Subjects receiving treatment with one or more drugs listed in the prohibited medication section.
* Regular use of oral or systemic corticosteroids for diseases other than asthma within the past 12 months or any intra-articular or short-acting, intramuscular corticosteroid within 1 month or intramuscular, long-acting depot corticosteroids within 3 months prior to screening.
* Subjects with severe hepatitis chronic active hepatitis or evidence of uncontrolled chronic liver disease.
* Subjects with Alanine Aminotransferase (ALT) or Aspartate Aminotransferase (AST) at screening ≥2x Upper Limit of Normal.
* Subjects with other severe acute or chronic medical or malignancy or psychiatric conditions which are uncontrolled or laboratory abnormality that may increase the risk associated with study participation or study drug administration or may interfere with the interpretation of study results and, would make the subjects inappropriate for entry into this study.
* Subjects with a history of lung volume resection.
* Subjects with a diagnosis of lung cancer or a history of lung cancer.
* Subjects with active cancer or a history of cancer (other than lung) with less than 5 years disease free survival time (whether or not there is evidence of local recurrence or metastases). Localised carcinoma (e.g. basal cell carcinoma, in situ carcinoma of the cervix adequately treated) is acceptable.
* Subjects who have received an investigational drug within 30 days (60 days for biologics) or five half-lives (whichever is greater) prior to screening visit.
* Subjects with a history of alcohol or drug abuse within two years prior to screening visit.
* Subjects with major surgery in the 3 months prior to screening visit or planned surgery during the trial.
* Subjects mentally or legally incapacitated or subjects accommodated in an establishment as a result of an official or judicial order.

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 810 (Actual)
Dates: Start 2019-08-28 (Actual); Primary Completion 2020-10-19 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
Efficacy of CHF 6532 on moderate and severe asthma exacerbations rate | Over 52 weeks of treatment
  Rate of moderate and severe asthma exacerbations during the treatment period with CH 6532 (3 doses tested) or Placebo

SECONDARY OUTCOMES:
Effect of CHF 6532 on severe asthma exacerbations compared to Placebo | Over 52 weeks of treatment
  Assessment of time to first moderate or severe exacerbation, and of time to first severe exacerbation
Effect of CHF 6532 compared to Placebo in terms of change from baseline in pre-dose morning FEV1 (Forced Expiratory Volume in 1 second) | At Week 52
  Assessment of change from Baseline in pre-dose FEV1
Effect of CHF 6532 compared to Placebo in terms of change from baseline on St. George's Respiratory Questionnaire (SGRQ) | At Week 52
  Assessment of change from Baseline in SGRQ scores (Score range from 0 to 100, with lower scores corresponding to better health)
Effect of CHF 6532 compared to Placebo in terms of change from baseline on Asthma Control Questionnaire (ACQ-5) | At Week 52
  Assessment of change from Baseline in ACQ-5 scores (Score range from 0=no impairment to 6= maximum impairment)
Effect of CHF 6532 compared to Placebo in terms of change from baseline on Asthma Quality of Life Questionnaire (AQLQ+12) | At Week 52
  Assessment of change from Baseline in AQLQ+12 scores (Score range from 1=severe impairment to 7= no impairment)
Pharmacokinetic analysis of CHF 6532 | At baseline and 3 months
  Assessment of the area Under of the plasma concentration-time curve from 0 to the last quantifiable concentration (AUC0-t) of CHF 6532
Pharmacokinetic analysis of CHF 6532 | At baseline and 3 months
  Assessment of the area Under of the plasma concentration versus time curve observed from time 0 up to 8 hours post-dose (AUC0-8h) of CHF 6532
Pharmacokinetic analysis of CHF 6532 | At baseline and 3 months
  Assessment of the value of the maximum plasma concentration (Cmax) of CHF 6532
Pharmacokinetic analysis of CHF 6532 | At baseline and 3 months
  Assessment of the time of the maximum plasma concentration (tmax) of CHF 6532

CONTACTS AND LOCATIONS:
Overall Officials: Pierluigi Paggiaro, MD, Principal Investigator — Universita di Pisa, Italy
Locations (1):
- Medical Center "Nov Rehabilitatsionen Tsentar" Ltd, Stara Zagora, Bulgaria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Study Record on EU Clinical Trials Register including results — https://www.clinicaltrialsregister.eu/ctr-search/trial/2018-003548-22/results
- See also: Lay Summaries of study results available in the CHIESI Clinical Study Register — https://www.chiesi.com/en/chiesi-clinical-study-register/